CLINICAL TRIAL: NCT02690051
Title: BeSmooth Study, a Physician-initiated PMCF Trial Investigating the BeSmooth Peripheral Stent System for the Treatment of Iliac Lesions
Brief Title: BeSmooth Study, Investigating the BeSmooth Peripheral Stent System for the Treatment of Iliac Lesions
Acronym: BeSmooth
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Flanders Medical Research Program (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMRP-140702
Record Dates: First submitted 2016-02-02; First posted 2016-02-24 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-02

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BeSmooth Peripheral Stent system (Experimental): Patients treated with the BeSmooth Peripheral Stent System
  Interventions: Device: BeSmooth peripheral stent

INTERVENTIONS:
Device: BeSmooth peripheral stent — patients treated with the BeSmooth Peripheral Stent System

SUMMARY:
A Physician initiated PMCF Trial Investigating the BeSmooth Peripheral Stent System for the treatment of Iliac Lesions.

The objective of this clinical investigation is to evaluate the long-term safety and efficacy of the BeSmooth Peripheral Stent System in clinical settings post CE-certification when used according to the indications of the IFU.

ELIGIBILITY:
Inclusion Criteria:

1. Corresponding to the CE-mark indications/contra-indications and according to the current medical guidelines for minimally invasive peripheral interventions.
2. Patient presenting with a stenotic or occlusive lesion at the iliac arteries suitable for stenting (on indication for primary stenting, based on the discretion of the investigator)
3. Patient presenting a score from 2 to 5 following Rutherford classification
4. Patient is willing to comply with specified follow-up evaluations at the specified times for the duration of the study
5. Patient is >18 years old
6. Patient (or their legal representative) understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
7. Patient is eligible for treatment with the BeGraft Peripheral Stent Graft System (Bentley InnoMed)
8. The target lesion is either a modified TASC-II class A, B, C or D lesion with one of the listed specifications:

   * Type A lesions

     * Unilateral or bilateral stenoses of the Common Iliac Artery
     * Unilateral or bilateral single short (≤3 cm) stenosis of the External Iliac Artery
   * Type B lesions

     * Unilateral Common Iliac Artery occlusion
     * Single or multiple stenosis totaling 3-10 cm involving the External Iliac Artery not extending into the Common Femoral Artery
     * Unilateral External Iliac Artery occlusion not involving the origins of Internal Iliac Artery or Common Iliac Artery
   * Type C lesions

     * Bilateral Common Iliac Artery occlusions
     * Bilateral External Iliac Artery stenoses 3-10 cm long not extending into the Common Femoral Artery
9. The target lesion has angiographic evidence of stenosis or restenosis > 50% or occlusion which can be passed with standard guidewire manipulation
10. There is angiographic evidence of a patent Common an Deep Femoral Artery

Exclusion Criteria:

1. PTA is technically not possible (not feasible to access the lesion or a defect with the guidewire or balloon catheter)
2. Presence of an aneurysm immediately adjacent to the site of stent implantation
3. Stenosis distal to the site of stent implantation
4. Lesions in or adjacent to essential collaterals(s)
5. Lesions in locations subject to external compression
6. Heavily calcified lesions resistant to PTA
7. Patients with diffuse distal disease resulting in poor stent outflow
8. Patients with a history of coagulation disorders
9. Patients with aspirin allergy or bleeding complications and patients unable or unwilling to tolerate anticoagulant/antiplatelet therapy and/or non-responders to anticoagulant/antiplatelet therapy
10. Fresh thrombus formation
11. Patients with known hypersensitivity to the stent material(L605)
12. The target lesion is either a modified TASC-II class B or D lesion with aortic or common femoral lesion involvement:

    * Type B lesions

      -Short (≤3 cm) stenosis of infrarenal aorta
    * Type C lesions

      * Unilateral External Iliac Artery stenosis extending into the Common Femoral Artery
      * Unilateral External Iliac Artery occlusion that involves the origins of the Internal Iliac and/or Common Femoral Artery
      * Heavily calcified unilateral External Iliac Artery occlusion with or without involvement of origins of the Internal Iliac and/or Common Femoral Artery
    * Type D lesions

      * Infra-renal aortoiliac occlusion
      * Iliac stenoses in patients with an Abdominal Aortic Aneurysm (AAA) requiring treatment and not amenable to endograft placement or other lesions requiring open aortic or iliac surgery
      * Diffuse multiple stenoses involving the unilateral Common Iliac, External Iliac and Common Femoral Artery
      * Unilateral occlusions of both Common Iliac and External Iliac Artery
      * Diffuse disease involving the aorta and both iliac arteries requiring treatment
      * Bilateral occlusions of the External Iliac Artery
13. Previously implanted stent(s) at the same lesion site
14. Reference segment diameter is not suitable for the available stent design
15. Untreatable lesion located at the distal outflow arteries
16. Use of alternative therapy (e.g. atherectomy, cutting balloon, laser, radiation therapy) as part of the index procedure
17. Patients refusing treatment
18. Patients for whom antiplatelet therapy, anticoagulants or thrombolytic drugs are contraindicated
19. Patients who exhibit persistent acute intraluminal thrombus of the proposed lesion site
20. Perforation at the angioplasty site evidenced by extravasation of contrast medium
21. Patients with a history of prior life-threatening contrast medium reaction
22. Patients with uncorrected bleeding disorders
23. Female patient with child bearing potential not taking adequate contraceptives or currently breastfeeding
24. Life expectancy of less than twelve months
25. Any planned surgical intervention/procedure within 30 days of the study procedure
26. Any patient considered to be hemodynamically unstable at onset of procedure
27. Patient is currently participating in another investigational drug or device study that has not completed the entire follow up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Primary Patency at 12 months | 12 months
  defined as a target lesion without a hemodynamically significant stenosis on duplex ultrasound (>50%, systolic velocity ratio no greater than 2.4) and without Target Lesion Revascularization (TLR) within 12 months.

SECONDARY OUTCOMES:
Primary Patency at 1 & 6 month | 1 and 6 months
  Patients that present without a hemodynamically significant stenosis at the target area on duplex ultrasound (>50%, systolic velocity ratio no greater than 2.4) and without prior TLR are defined as being primary patent at the given follow-up.
Stent Occlusion Rate at 1,6 and 12-month follow-up | up to 12 months
  100% (re)occlusion rate within the study stent
ABI at 1,6 and 12-month follow-up, compared with baseline | up to 12 months
  Ankle-Brachial index measurements at 1,6 and 12-month FU visit, compared with measurements at baseline (pre operatively)
Amputation rate at 1,6 and 12-month follow-up | up to 12 months
  Amputation rate at 1-, 6- and 12-month follow-up, defined as any amputation above the knee.
Performance success rate at baseline, defined as restoration of blood flow | during the index study procedure
  Device success, restoration of blood flow during index procedure
In-stent restenosis rate | up to 12 months
  restenosis rate within the study stent
Freedom from Target Lesion Revascularization | up to 12 months
  Freedom from Target Lesion Revascularization (TLR), defined as freedom from a repeat intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5mm proximal and distal to the treated lesion edge.
Serious Adverse Events | up to 12 months
  Serious Adverse Events (SAEs), defined according to ISO 14155:2011 as any clinical event that is fatal, life-threatening, or judged to be severe by the investigator; resulted in persistent or significant disability; necessitated surgical or percutaneous intervention; or required prolonged hospitalization.
Technical success | during the index study procedure
  The ability to achieve final residual angiographic stenosis no greater than 30%
Clinical success at follow-up is defined as an improvement of Rutherford Classification at 1-,6- and 12-month follow-up | up to 12 months
  Clinical success at follow-up is defined as an improvement of Rutherford classification at 1-, 6- and 12-month follow-up of one class or more as compared to the pre-procedure Rutherford classification

CONTACTS AND LOCATIONS:
Overall Officials: Koen Deloose, MD, Principal Investigator — Flanders Medical Research Program
Locations (4):
- Belgium (4):
  - OLV Hospital, Aalst
  - Imelda Hospital Bonheiden, Bonheiden
  - AZ Sint-Blasius, Dendermonde
  - Heilig Hart Hospital, Tienen

IPD SHARING:
Plan to Share IPD: Undecided